CLINICAL TRIAL: NCT07202533
Title: Investigation of the Effectiveness of Exercise and Pain Neuroscience Education in Individuals With Chronic Nonspecific Low Back Pain With Central Sensitization
Brief Title: Pain Neuroscience Education and Exercise for Chronic Nonspecific Low Back Pain
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ayşe ŞİMŞEK, → PhD Candidate, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Hacettepe-FTR-AŞ-01
Record Dates: First submitted 2025-09-02; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Chronic Non-specific Low Back Pain
Keywords: low back pain; central sensitization; surface electromyography; pain neuroscience education; motor control exercise
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either a control group receiving motor control exercises or an intervention group receiving motor control exercises plus PNE. Both groups will receive treatment twice weekly for 8 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motor Control Exercises (Active Comparator): This group will receive motor control exercises only.
  Interventions: Other: Motor Control Exercises
- Motor Control Exercises + Pain Neuroscience Education (Experimental): This group will receive the same motor control exercise program as the control group, plus a 6-week PNE program delivered once per week. The PNE program consists of 6 weekly sessions, delivered via slide presentations and interactive discussions, covering topics such as nociception, central sensitization, neuroplasticity, and pain coping strategies. Sessions are delivered by a certified physiotherapist.
  Interventions: Other: Pain Neuroscience Education; Other: Motor Control Exercises

INTERVENTIONS:
Other: Motor Control Exercises — Participants will perform these exercises under physiotherapist supervision twice per week for 8 weeks. Exercises focus on improving deep trunk muscle coordination and stability.
  Arms: Motor Control Exercises
Other: Pain Neuroscience Education — A 6-week educational program with weekly sessions using slide presentations and interactive discussions, covering pain neurophysiology, central sensitization, and pain coping strategies, delivered by a certified physiotherapist.
  Arms: Motor Control Exercises + Pain Neuroscience Education
Other: Motor Control Exercises — Participants will perform these exercises under physiotherapist supervision twice per week for 8 weeks. Exercises focus on improving deep trunk muscle coordination and stability.
  Arms: Motor Control Exercises + Pain Neuroscience Education

SUMMARY:
This study aims to evaluate the effects of adding Pain Neuroscience Education (PNE) to motor control exercises in individuals with chronic non-specific low back pain (CNSLBP) who also present with central sensitization. The study focuses on changes in pain intensity, pain-related factors, trunk muscle activation, gait, functionality, kinesiophobia, and quality of life.

DETAILED DESCRIPTION:
This randomized controlled study aims to investigate the effects of combining PNE with motor control exercises in individuals with CNSLBP who demonstrate central sensitization (≥28 points on the Central Sensitization Inventory). Participants are randomly assigned into two groups: the intervention group (motor control exercises + PNE) and the control group (motor control exercises only). Both groups participate in motor control exercises twice a week for 8 weeks, under the supervision of a physiotherapist. The intervention group additionally receives six PNE sessions once per week for six weeks. PNE sessions are delivered by a certified physiotherapist using interactive presentations and question-answer discussions.

Assessments are performed pre- and post-intervention using the following tools:

* Central Sensitization Inventory (CSI) to determine the presence and severity of central sensitization.
* Numeric Pain Rating Scale (NPRS) for pain intensity.
* Revised Neurophysiology of Pain Questionnaire (rNPQ) for pain knowledge.
* Pain Catastrophizing Scale (PCS) for catastrophic thinking.
* Pressure Pain Threshold (PPT) using a digital algometer.
* Electromyographic (EMG) evaluation of trunk and lower extremity muscles using surface electrodes.
* Spatiotemporal gait analysis using OptoGait and Ultium Insole systems.
* Tampa Scale for Kinesiophobia (TSK) for fear of movement.
* Roland-Morris Disability Questionnaire (RMDQ) for disability level.
* Nottingham Health Profile (NHP) for quality of life.

Data will be analyzed using SPSS version 27. Normality of distribution will be tested with the Shapiro-Wilk test. Depending on the distribution, either parametric (paired t-test, independent t-test) or non-parametric tests (Wilcoxon signed-rank, Mann-Whitney U) will be applied. Pearson or Spearman correlation analyses will be used where appropriate.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers who agree to participate in the study
* Having a history of non-specific low back pain lasting at least 3 months
* Having a pain intensity score of 3 or higher on the Numerical Pain Rating Scale (NPRS) within the last week
* Scoring ≥28 on the Turkish version of the Central Sensitization Inventory.

Exclusion Criteria:

* Individuals with radicular symptoms or cauda equina syndrome
* Severe osteoporosis
* Spondyloarthropathy
* Spondylolisthesis
* Lumbar spinal stenosis
* Lumbar fractures
* Malignant tumors
* Severe comorbidities (neurological, neuromuscular, cardiac, or psychiatric disorders)
* Individuals who have undergone spinal surgery
* Individuals who are familiar with motor control exercises or who have previously received pain neuroscience education

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-29 (Actual); Primary Completion 2025-08-08 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity (Numerical Pain Rating Scale - NPRS) | Baseline and post-intervention (8 weeks)
  Change in pain intensity will be assessed using a 0-10 Numerical Pain Rating Scale at baseline and post-intervention. Higher scores indicate greater pain severity.
Pressure Paın Threshold Measurement | Baseline and post-intervention (8 weeks)
  PPT will be measured using a digital algometer on the lumbar region. Higher values indicate reduced pain sensitivity.
Central Sensitization (Central Sensitization Inventory - CSI) | Baseline and post-intervention (8 weeks)
  The CSI-A section will be used to evaluate symptoms related to central sensitization. Total scores range from 0-100, with higher scores indicating greater sensitization.
Pain Knowledge (Revised Neurophysiology of Pain Questionnaire - rNPQ) | Baseline and post-intervention (8 weeks)
  Participants' knowledge about pain neurophysiology will be assessed. The number of correct responses will be calculated.
Disability (Roland-Morris Disability Questionnaire - RMDQ) | Baseline and post-intervention (8 weeks)
  Functional disability due to low back pain will be assessed using the RMDQ, a 24-item self-report questionnaire.
Muscle Activation (Surface EMG Analysis) | Baseline and post-intervention (8 weeks)
  Surface EMG will evaluate activation levels of bilateral external oblique, internal oblique, transversus abdominis, and tibialis anterior muscles during gait.

SECONDARY OUTCOMES:
Kinesiophobia (Tampa Scale for Kinesiophobia - TSK) | Baseline and post-intervention (8 weeks)
  Fear of movement will be evaluated with the TSK. Total scores range from 17-68. Higher scores represent more fear-avoidance behavior.
Pain Catastrophizing (Pain Catastrophizing Scale - PCS) | Baseline and post-intervention (8 weeks)
  Total PCS scores will be used to assess exaggerated negative thoughts related to pain. Higher scores indicate greater catastrophizing.
Gait Analysis (OptoGait Photocell System) | Baseline and post-intervention (8 weeks)
  Spatiotemporal characteristics of gait will be assessed using a validated and reliable treadmill-based OptoGait photocell system (Version 1.6.4.0, Microgate, Bolzano, Italy). All participants will be asked to walk on the treadmill and select a speed at which they feel most comfortable. After the participant has become accustomed to walking on the treadmill and determined their preferred speed, spatiotemporal parameters will be recorded during a one-minute walking trial.
Gait Analysis (Noraxon Ultium Insole) | Baseline and post-intervention (8 weeks)
  Spatiotemporal gait parameters will be assessed using the Ultium Insole SmartLead pedobarographic analysis system (SmartLead, Noraxon, Scottsdale, AZ, USA). Participants will walk at a self-selected comfortable speed in a controlled laboratory environment, and each will perform the walking task three times. Data will be collected via Noraxon software during overground walking, including stance phase percentage, swing phase percentage, step duration (ms), double support duration (ms), and cadence (steps/min).
Quality of Life (Nottingham Health Profile - NHP) | Baseline and post-intervention (8 weeks)
  Quality of life will be evaluated using the Nottingham Health Profile, covering six dimensions: physical mobility, pain, sleep, energy, social isolation, and emotional reactions.

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Ankara, Karabük Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No